CLINICAL TRIAL: NCT04691492
Title: Harnessing the Power of Friends to Reduce Alcohol-Involved Sexual Assault Risk
Brief Title: Protecting Allies in Risky Situations
Acronym: PAIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jennifer Read, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34AA027046 (NIH); R34AA027046 (NIH)
Record Dates: First submitted 2020-12-11; First posted 2020-12-31 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Sexual Assault; College Drinking; Behavioral Changes
MeSH Terms: conditions — Alcohol Drinking in College

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Friends-Based Motivational Interview (FMI) Group (Experimental): Will participate in the Friends-Based Motivational Interview (FMI) program.
  Interventions: Behavioral: Friend-Based Motivational Interview
- Wait List Control (No Intervention): The Wait List Control group will also be offered to participate in the Friends-Based Motivational Interview Program but at a deferred date (12 weeks later).

INTERVENTIONS:
Behavioral: Friend-Based Motivational Interview — The intervention will use Motivational Interviewing's (MI) collaborative conversation style for strengthening commitment to change, to motivate and prepare women to work together to reduce Sexual Assault (SA) risk. This intervention will target ways that the friend dyad may support, encourage, and share responsibility with one another in protecting against SA. The Friend-based MI (FMI) will then use the responsibility and relationship of friends as a framework to foster collaborative efforts to increase readiness and decrease barriers to helping behavior. As part of this, the FMI will focus on the identification and implementation of skills friends can use to help one another prevent sexual assault. FMI will include a focused discussion of the ways drinking may impede helping efforts. Moreover, the FMI will encourage women to identify personal, specific strategies for reducing the effects of alcohol on helping.
  Arms: Friends-Based Motivational Interview (FMI) Group

SUMMARY:
The current project will provide testing of a friend-based motivational interview (FMI) designed to reduce sexual assault risk. The study will address if the intervention minimizes the impact of alcohol on helping behavior, test whether drinking reduces intervention efficacy, and examine potential iatrogenic effects of the intervention.

DETAILED DESCRIPTION:
The objective of the proposed study is to develop an innovative, friend-based motivational interview (FMI) that encourages and prepares friends to reduce sexual assault (SA) risk. Delivered to pairs of friends (dyads), the FMI will be designed to foster collaborative efforts to increase readiness for, and decrease barriers to helping behavior, and to teach and plan together for assault prevention skills. As the role of alcohol has been under-addressed in SA prevention efforts, the FMI also will explicitly attend to how intoxication may serve as a barrier to friend intervention, and strategies for overcoming this barrier. The completion of this project's aims will yield a novel intervention that capitalizes on the natural resource of women's friendships to decrease risk for sexual assault - a pervasive public health problem affecting a substantial portion of young adult women in the U.S.

Twenty-four friend dyads will participate in the friend-based motivational interview (FMI) along with 24 wait-list control dyads (total of 48 dyads). The study will compare groups on outcomes at post-intervention and at bi-weekly 3 month follow-ups, and also examine within participant change. The study will focus on whether effects are in the expected direction and whether the strength of effect sizes are of practical magnitude. It is expected that participants receiving the FMI will demonstrate significant increases in readiness, and engagement in friend assault prevention behavioral skills (FAPBs), and demonstrate decreases in perceived barriers, at post-intervention and over the 3-month follow-up. Follow-up data will be utilized to provide a rich description of the role of alcohol in implementing FAPBs, and whether the FMI reduces the impact of alcohol use. In exploratory analyses, it will be examined whether the intervention may be associated with decreased assault risk, as well as decreased drinking.

ELIGIBILITY:
Inclusion Criteria:

* Female dyads who go out together at least once a week
* Undergraduates enrolled in a 4-year college or university
* Meet heavy episodic drinking (HED) criteria, 4 or more drinks in a single sitting, 2 or more times monthly

Exclusion Criteria:

Not Applicable

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer P Read, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo Department of Psychology, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share a de-identified data set which will include baseline demographics and readiness to intervene, awareness of alcohol's effects on helping behaviors, friend-based assault protective strategy use, and perception of barriers to intervening outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available in December 2021 and will be available until 2026.
Access Criteria: There must be an articulation of a clear research question and analytic plan by an established investigator with the relevant credentials. The information will be shared as a digital file through email.

REFERENCES:
- [Derived] Read JP, Livingston JA, Shaw RJ, Wiseblatt AF, Jenzer T, DiPaolo LR, Mastroleo NR, Katz J, Testa M, Colder CR. The power of friends in reducing sexual assault risk in college women: A preliminary test of dyad-based motivational intervention approach. J Consult Clin Psychol. 2024 Dec;92(12):814-827. doi: 10.1037/ccp0000925. PMID 39715424

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (N=108, 54 dyads) were recruited using a multi-method, community-based recruitment plan, including: digital and print advertisements, social media, email blasts to psychology and nursing student listservs, flyers posted in locations frequented by emerging adults (e.g., college campuses, coffee shops, bars) and word of mouth. A QR code and/or link directed interested individuals to a secure platform to learn more about the trial and complete a brief initial eligibility questionnaire.
Period: Overall Study
Arm/Group | Friends-Based Motivational Interview (FMI) Group | Wait List Control
Started | 56 | 52
Completed | 50 | 52
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Population: 6 participants dropped out before completing the baseline which is why the total here is 102 where the total enrollment was 108.
Groups:
- Total: Total of all reporting groups
Arm/Group | Friends-Based Motivational Interview (FMI) Group | Wait List Control | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 52 | 102
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.62 (1.01) | 19.48 (1.06) | 19.6 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 52 | 102
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 3 | 8
  White | 35 | 34 | 69
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 50 | 52 | 102
Year in College [Count of Participants; unit: Participants]
  Freshman | 8 | 6 | 14
  Sophomore | 15 | 25 | 40
  Junior | 15 | 13 | 28
  Senior | 12 | 8 | 20
Housing [Count of Participants; unit: Participants]
  Residence Hall | 17 | 19 | 36
  On campus | 4 | 7 | 11
  Home (with family) | 6 | 6 | 12
  House or apartment (off campus, not with family) | 23 | 20 | 43
GPA [Mean (Standard Deviation); unit: units on a scale] — Grade Point Average (GPA) is 4 point scale used by most colleges to average the grades of students. The range is 0.0-4.0 with a 4.0 representing higher grades on average. The score is obtained by converting each letter grade a student received into a number (A=4, A-=3.67, B+=3.33, B=3...) then finding the mean of those numbers.
  units on a scale | 3.30 (0.47) | 3.28 (0.51) | 3.29 (0.49)
Greek Affiliation [Count of Participants; unit: Participants]
  No | 43 | 42 | 85
  Yes | 7 | 10 | 17
Employed [Count of Participants; unit: Participants]
  No, I'm not working | 18 | 25 | 43
  Yes, part time (irregular hours) | 25 | 12 | 37
  Yes, part-time (approximately 20 hours) | 6 | 12 | 18
  Yes, full-time (approximately 40 hours) | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Readiness to Intervene on the Readiness Ruler
Description: Participants will use an 11-point likert-type scale modeled after the Readiness Ruler to rate their readiness for intervening. Responses range from 0 (I never think about my and/or my friend's risk of being sexually assaulted) to 10 (I am actively and consistently taking steps to protect myself and/or my friends from sexual assault), with higher scores indicating a greater readiness to intervene.
Time Frame: Baseline and Monthly for 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friends-Based Motivational Interview (FMI) Group | Wait List Control
Number analyzed (Participants) | 50 | 52
score on a scale
  Baseline | 7.22 (1.74) | 7.44 (1.97)
  Month 1 | 8.60 (2.19) | 7.29 (1.71)
  Month 2 | 8.52 (1.15) | 7.50 (1.59)
  Month 3 | 9.15 (0.9) | 7.77 (1.68)

2. Primary Outcome: Change in Readiness to Intervene on the Decisional Balance Scale
Description: The 10-item Decisional Balance Scale (Banyard et al., 2007) is used to assess ambivalence about intervening in a potential assault situation. Responses regarding the decision whether to intervene or not are rated on a 5-point Likert scale ranging from 1 (Not at all likely) to 5 (Extremely likely), with higher scores indicating a greater readiness to intervene.
Time Frame: Baseline and 3 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friends-Based Motivational Interview (FMI) Group | Wait List Control
Number analyzed (Participants) | 50 | 52
score on a scale
  Baseline | 4.92 (0.13) | 4.94 (0.14)
  Month 3 | 4.86 (0.41) | 4.83 (0.38)

3. Primary Outcome: Change in Awareness and Strategies Regarding Alcohol Effects on Helping Survey
Description: This 8-item survey measures awareness of and strategies for alcohol's effects on helping behavior and participants' understanding of the ways that alcohol may interfere with helping behavior. Responses range from 1 (Not at all true) to 5 (Very much true), with higher scores indicating a greater understanding of how alcohol interferes with helping behavior.
Time Frame: Baseline and Monthly for 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friends-Based Motivational Interview (FMI) Group | Wait List Control
Number analyzed (Participants) | 50 | 52
score on a scale
  Baseline | 2.75 (0.61) | 2.66 (0.59)
  Month 1 | 2.81 (0.68) | 2.73 (0.59)
  Month 2 | 2.66 (0.69) | 2.65 (0.68)
  Month 3 | 2.73 (0.63) | 2.54 (0.90)

4. Primary Outcome: Change in Friend-Based Helping Skills on Friend-based Assault Protective Strategies Assessment
Description: The Friend-based Assault Protective Strategies Assessment uses 20 items to assess sexual assault preventive strategy use. Responses range from 1 (Not at all) to 4 (A lot), with higher scores indicating a greater use of strategies to prevent sexual assault.
Time Frame: Baseline and Monthly for 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friends-Based Motivational Interview (FMI) Group | Wait List Control
Number analyzed (Participants) | 50 | 52
score on a scale
  Baseline | 1.98 (0.50) | 1.92 (0.51)
  Month 1 | 2.19 (0.60) | 1.88 (0.63)
  Month 2 | 1.95 (0.65) | 1.97 (0.65)
  Month 3 | 2.45 (0.51) | 1.90 (0.62)

5. Primary Outcome: Change in Friend-Based Helping Skills on the Bystander Behaviors Scale for Friends
Description: We used a modified version of The Bystander Behaviors Scale for Friends is a 44-item measure which includes 4 sub-scales (1) the identification of sexual assault risk situations, (2) accessing resources, (3) planning ahead for risk situations, and (4) safety behaviors in risk settings. We used a selection of 20 questions from the full measure including items from each subscale. Response option include (0) No I did not engage in this behavior, (1) Yes I did engage in this behavior, or (missing) I did not perceive an opportunity to engage in this behavior. A higher endorsement of "Yes" (higher score) engaging in the behaviors is considered to indicate a greater use of strategies to prevent sexual assault.
Time Frame: Baseline and Monthly for 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friends-Based Motivational Interview (FMI) Group | Wait List Control
Number analyzed (Participants) | 50 | 52
score on a scale
  Baseline | 0.86 (0.18) | 0.87 (0.19)
  Month 1 | 0.89 (0.23) | 0.83 (0.25)
  Month 2 | 0.80 (0.35) | 0.78 (0.28)
  Month 3 | 0.88 (0.26) | 0.82 (0.29)

6. Primary Outcome: Change in Perceived Barriers to Intervening on the Barriers to Sexual Assault Bystander Intervention Scale
Description: The Barriers to Sexual Assault Bystander Intervention Scale is a 16-item measure to assess barriers to intervening. Responses range from 1 (Strongly disagree) to 7 (Strongly agree), with higher scores indicating greater perceived barriers to intervening.
Time Frame: Baseline and Monthly for 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friends-Based Motivational Interview (FMI) Group | Wait List Control
Number analyzed (Participants) | 50 | 52
score on a scale
  Baseline | 2.43 (0.80) | 2.39 (0.76)
  Month 1 | 2.57 (0.89) | 2.57 (0.87)
  Month 2 | 2.47 (0.89) | 2.53 (0.93)
  Month 3 | 2.39 (0.94) | 2.47 (0.89)

7. Primary Outcome: Change in Perceived Barriers to Intervening on the Concerns About Intervening Scale
Description: The Concerns About Intervening Scale uses 6 items to assess perceived barriers to intervening, focused on worries. Responses range from 1 (Not at all true) to 6 (Very much true), with higher scores indicating greater perceived barriers to intervening.
Time Frame: Baseline and Monthly for 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friends-Based Motivational Interview (FMI) Group | Wait List Control
Number analyzed (Participants) | 50 | 52
score on a scale
  Baseline | 1.81 (0.72) | 1.81 (0.62)
  Month 1 | 2.01 (0.85) | 1.95 (0.72)
  Month 2 | 1.97 (0.87) | 1.80 (0.75)
  Month 3 | 1.88 (0.84) | 1.93 (0.76)

8. Secondary Outcome: Sexual Assault
Description: Revised Sexual Experiences Survey (R-SES) will be used to assess each social occasion with the target friend in the prior 2 weeks. Each item will be coded 1 (yes) or 0 (no), based on whether it happened to the woman/friend on each occasion that the pair socialized together.
Time Frame: Monthly after baseline for 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Friends-Based Motivational Interview (FMI) Group | Wait List Control
Number analyzed (Participants) | 50 | 52
Participants
  Month 1: No | 44 | 42
  Month 1: Yes | 2 | 5
  Month 1: Prefer not to answer | 4 | 5
  Month 2: No | 45 | 43
  Month 2: Yes | 2 | 5
  Month 2: Prefer not to answer | 3 | 4
  Month 3: No | 46 | 50
  Month 3: Yes | 1 | 0
  Month 3: Prefer not to answer | 3 | 2

9. Secondary Outcome: Change in Drinking
Description: Using a grid-based average assessment measure based in the Daily Drinking Questionnaire, participants will report on alcohol consumption. Higher scores indicate greater alcohol consumption.
Time Frame: Baseline and Monthly for 3 months
Measure: Mean (Standard Deviation); unit: Amount of drinks consumed weekly
Arm/Group | Friends-Based Motivational Interview (FMI) Group | Wait List Control
Number analyzed (Participants) | 50 | 52
Amount of drinks consumed weekly
  Baseline | 9.84 (5.34) | 10.79 (7.93)
  Month 1 | 7.06 (4.96) | 8.92 (4.77)
  Month 2 | 6.13 (7.13) | 7.38 (6.14)
  Month 3 | 6.27 (6.32) | 7.77 (6.15)

ADVERSE EVENTS:
Time Frame: No assessment after the conclusion of data collection. So at baseline, biweekly for 12 weeks for treatment and monthly for 3 months for waitlist.
Arm/Group | Friends-Based Motivational Interview (FMI) Group | Wait List Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/52
Other Adverse Events (participants affected / at risk) | 0/50 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT04691492/Prot_SAP_000.pdf